CLINICAL TRIAL: NCT04409626
Title: Is Hyponatraemia a Risk Factor for Mortality in Schizophrenic and Bipolar Patients? Protocol for a Bayesian Causal Inference Study
Brief Title: Hyponatraemia and Mortality in Schizophrenic and Bipolar Patients: Protocol for a Bayesian Causal Inference Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-2020-05-05
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Hyponatremia; SIADH
Keywords: Causality; Bayesian analysis; Antipsychotics; Psychotropics; Polypharmacy
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases
  Interventions: Other: Plasma sodium level (continuous variables)
- Controls: Matched (5 controls per case) by date of birth +/- 180 days.
  Interventions: Other: Plasma sodium level (continuous variables)

INTERVENTIONS:
Other: Plasma sodium level (continuous variables) — Observational study, so the exposures of interest (5-year mean and minimum plasma sodium) are not administered to the patients. Ultimately, our interest is in hyponatraemia.

SUMMARY:
This study seeks to investigate if hyponatraemia be a direct contributor to death in schizophrenic and bipolar patients, and gauge the potential role of somatic comorbidity and psychotropic polypharmacy, with emphasis on antipsychotics and antidepressants.

ELIGIBILITY:
Source population:

* Danish residents
* At least one International Classification of Diseases version 10 (ICD-10) F2 or F31 diagnosis from a hospital in Region Zealand and the Capital Region (Denmark)

No exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases:
  * Died in our catchment area between 1 January 2011 and 1 July 2016.
  Controls:
  * 5 controls per case found by risk-set sampling with replacement, matched on date of birth +/- 180 days.
Sampling Method: Probability Sample
Enrollment: 31740 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 January 2011 through 1 July 2016
  All-cause mortality

IPD SHARING:
Plan to Share IPD: No
We are unfortunately unable to share individual participant data, as our data source comprises sensitive information from electronic medical records and national registries.